CLINICAL TRIAL: NCT00945698
Title: A Two-centre, Randomised, Single-blind, Parallel Group Controlled Trial, Testing the Growth Promoting Effect of Long-term Complementary Feeding of Infants With Different Doses and Formulations of Lipid-based Nutrient Supplements (LNS)
Brief Title: Prevention of Linear Growth Failure in Infants and Young Children With Lipid-based Nutrient Supplements (iLiNS-DOSE)
Acronym: iLiNS-DOSE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tampere University (Other)
Collaborators: Kamuzu University of Health Sciences (Other); University of California, Davis (Other); Bill and Melinda Gates Foundation (Other)
Responsible Party: Principal Investigator, Per Ashorn, Professor of International Health, Tampere University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: iLiNS-DOSE
Record Dates: First submitted 2009-07-21; First posted 2009-07-24 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2015-05

CONDITIONS: Malnutrition
Keywords: Stunting; Growth failure; Malnutrition; Lipid based nutrient supplement; LNS; Prevention; Malawi; Sub-Saharan Africa; Dietary supplementation; Efficacy
MeSH Terms: conditions — Malnutrition; Growth Disorders; Failure to Thrive

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- ST-DI (Delayed intervention) (Other): * 1 kg fortified maize / soy flour (Likuni phala, LP) 2-weekly (71 g / day) between 18 and 30 months of age
  * Normal under-five clinic follow-up, including EPI-vaccinations, vitamin A supplementation, and growth monitoring
  Interventions: Dietary Supplement: Maize-soy flour
- LNS-10gM (Experimental): * 140 g of milk-containing LNS (LNS-10gM) 2-weekly (10 g / day) between 6 and 18 months of age
  * Normal under-five clinic follow-up, including EPI-vaccinations, vitamin A supplementation, and growth monitoring
  Interventions: Dietary Supplement: Lipid-based nutrient supplement, 10gM
- LNS-20gM (Experimental): * 280 g of milk-containing LNS (LNS-20gM) 2-weekly (20 g / day) between 6 and 18 months of age
  * Normal under-five clinic follow-up, including EPI-vaccinations, vitamin A supplementation, and growth monitoring
  Interventions: Dietary Supplement: Lipid-based nutrient supplement, 20gM
- LNS-20gNoM (Experimental): * 280 g of milk-free LNS (LNS-20gNoM) 2-weekly (20 g / day) between 6 and 18 months of age
  * Normal under-five clinic follow-up, including EPI-vaccinations, vitamin A supplementation, and growth monitoring
  Interventions: Dietary Supplement: Lipid-based Nutrient Supplement, 20gNoM
- LNS-40gM (Experimental): * 560 g of milk-containing LNS (LNS-40gM) 2-weekly (40 g / day) between 6 and 18 months of age
  * Normal under-five clinic follow-up, including EPI-vaccinations, vitamin A supplementation, and growth monitoring
  Interventions: Dietary Supplement: Lipid-based nutrient supplement, 40gM
- LNS-40gNoM (Experimental): * 560 g of milk-free LNS (LNS-40gNoM) 2-weekly (40 g / day) between 6 and 18 months of age
  * Normal under-five clinic follow-up, including EPI-vaccinations, vitamin A supplementation, and growth monitoring
  Interventions: Dietary Supplement: Lipid-based Nutrient Supplement, 40gNoM

INTERVENTIONS:
Dietary Supplement: Lipid-based nutrient supplement, 10gM — * 140 g of milk-containing LNS (LNS-10gM) 2-weekly (10 g / day) between 6 and 18 months of age
  * Normal under-five clinic follow-up, including EPI-vaccinations, vitamin A supplementation, and growth monitoring
  Arms: LNS-10gM
Dietary Supplement: Lipid-based nutrient supplement, 20gM — * 280 g of milk-containing LNS (LNS-20gM) 2-weekly (20 g / day) between 6 and 18 months of age
  * Normal under-five clinic follow-up, including EPI-vaccinations, vitamin A supplementation, and growth monitoring
  Arms: LNS-20gM
Dietary Supplement: Lipid-based Nutrient Supplement, 20gNoM — * 280 g of milk-free LNS (LNS-20gNoM) 2-weekly (20 g / day) between 6 and 18 months of age
  * Normal under-five clinic follow-up, including EPI-vaccinations, vitamin A supplementation, and growth monitoring
  Arms: LNS-20gNoM
Dietary Supplement: Lipid-based nutrient supplement, 40gM — * 560 g of milk-containing LNS (LNS-40gM) 2-weekly (40 g / day) between 6 and 18 months of age
  * Normal under-five clinic follow-up, including EPI-vaccinations, vitamin A supplementation, and growth monitoring
  Arms: LNS-40gM
Dietary Supplement: Lipid-based Nutrient Supplement, 40gNoM — * 560 g of milk-free LNS (LNS-40gNoM) 2-weekly (40 g / day) between 6 and 18 months of age
  * Normal under-five clinic follow-up, including EPI-vaccinations, vitamin A supplementation, and growth monitoring
  Arms: LNS-40gNoM
Dietary Supplement: Maize-soy flour — * No food supplement during the primary trial period (6 to 18 months of age)
  * 1 kg fortified maize / soy flour (Likuni phala, LP) 2-weekly (71 g / day) between 18 and 30 months of age
  * Normal under-five clinic follow-up, including EPI-vaccinations, vitamin A supplementation, and growth monitoring
  Arms: ST-DI (Delayed intervention)

SUMMARY:
The use of lipid-based nutrients (LNS), such as Nutributter or fortified spread (FS), have been associated with improved growth and development outcomes among infants in Ghana and Malawi. Modified versions of such supplements have been developed to improve their nutrient density and quality and to lower their costs. Such modified products have proven acceptable to infants and their guardians in Malawi and Ghana. In the present trial, the investigator aim to identify the lowest growth-promoting daily dose of modified LNS. Additionally, the investigators will test a hypothesis that LNS that does not contain milk promotes growth as well as milk-containing LNS when given for 12 months at a 10-40 g daily dose to 6-18 month old infants in rural Malawi.

DETAILED DESCRIPTION:
Six-month old healthy infants are identified through community surveys in the study area. 1920 infants meeting set criteria are randomised into receiving the following intervention between 6 and 18 months of age: 1) standard treatment from 6-18 months (i.e.no supplements, with delayed intervention between 18-30 months of age (ST-DI), 2) 10 g / day milk-containing LNS (LNS-10gM), 3) 20 g / day milk-containing LNS (LNS-20gM), 4) 20 g / day milk-free LNS (LNS-20gNoM), 5) 40 g / day milk-containing LNS, (LNS-40gM) 6) 40 g / day milk-free LNS (LNS-40gNoM). The families receive the food supplements at 2-weekly intervals and the participants undergo a morbidity evaluation weekly, a limited development assessment at 4-weekly intervals and anthropometric evaluation at 26-week intervals and laboratory analyses at enrollment and at 18 months. Growth outcome analyses are done at 18 and at 42 months of age.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent from at least one guardian
* Age 5.50 months to 6.49 months
* Availability during the period of the study.
* Permanent resident of Mangochi District Hospital or Namwera Health Centre catchment area

Exclusion Criteria:

* Weight for length Z score (WLZ) < -2.0
* Presence of oedema
* Severe anaemia (Hb<50 g / l)
* Severe illness warranting hospital referral
* History of allergy towards peanut
* History of anaphylaxis or serious allergic reaction to any substance, requiring emergency medical care
* Concurrent participation in any other clinical trial

Ages: 167 Days to 197 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1920 (Estimated)
Dates: Start 2009-11; Primary Completion 2012-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Change in length-for-age Z-score (LAZ, based on WHO 2005 MGRS) between enrollment and 18 months of age | Primarily 12 months after enrollment (age 18 months), secondarily 36 months after enrollment (age 42 months)
Incidence of serious adverse events during the study period | 12 months after enrollment (age 18 months)

SECONDARY OUTCOMES:
Change in weight-for-age (WAZ) and weight-for-length (WLZ) Z-scores | Primarily 12 months after enrollment (age 18 months), secondarily 36 months after enrollment (age 42 months)
Incidence of stunting, underweight, and wasting | Primarily 12 months after enrollment (age 18 months), secondarily 36 months after enrollment (age 42 months)
Prevalence of reduced appetite | Daily assessment during 12 month supplementation
Energy intake from complementary foods | 3 and 9 months after enrollment (age 9 and 15 months)
Incidence of laboratory-confirmed malaria infection | 12 months after enrollment (age 18 months)
Incidence of caregiver-reported morbidity | Daily assessment during 12 month supplementation
Immune function (measured by humoral immunity towards measles vaccination) | 12 months after enrollment (age 18 months)
Change in hemoglobin and micronutrient status (iron status, measured by zinc protoporphyrin (ZPP); plasma zinc; plasma vitamin A; B-vitamins and related metabolites; urine iodine | 12 months after enrollment (age 18 months)
Proportion with anaemia at 18 months of age | 12 months after enrollment (age 18 months)
Change in erythrocyte essential fatty acid (EFA) concentration (measured from a subsample of 400 participants) | 12 months after enrollment (age 18 months)
Neuro-behavioral development (timing of acquisition of the certain skills and more comprehensive analysis at the age of 18 months) | Limited assessment every 4 weeks during the 12 months supplementation, more comprehensive at age 18 months
Incidence of all adverse events during the study period | 12 months after enrollment (age 18 months)

CONTACTS AND LOCATIONS:
Overall Officials: Per Ashorn, MD, PhD, Principal Investigator — University of Tampere Medical School; Kenneth Maleta, MBBS, PhD, Principal Investigator — Kamuzu University of Health Sciences
Locations (1):
- University of Malawi, College of Medicine, Mangochi, Malawi

REFERENCES:
- [Background] Adu-Afarwuah S, Lartey A, Brown KH, Zlotkin S, Briend A, Dewey KG. Home fortification of complementary foods with micronutrient supplements is well accepted and has positive effects on infant iron status in Ghana. Am J Clin Nutr. 2008 Apr;87(4):929-38. doi: 10.1093/ajcn/87.4.929. PMID 18400716
- [Background] Phuka JC, Maleta K, Thakwalakwa C, Cheung YB, Briend A, Manary MJ, Ashorn P. Complementary feeding with fortified spread and incidence of severe stunting in 6- to 18-month-old rural Malawians. Arch Pediatr Adolesc Med. 2008 Jul;162(7):619-26. doi: 10.1001/archpedi.162.7.619. PMID 18606932
- [Background] Phuka JC, Maleta K, Thakwalakwa C, Cheung YB, Briend A, Manary MJ, Ashorn P. Postintervention growth of Malawian children who received 12-mo dietary complementation with a lipid-based nutrient supplement or maize-soy flour. Am J Clin Nutr. 2009 Jan;89(1):382-90. doi: 10.3945/ajcn.2008.26483. Epub 2008 Dec 3. PMID 19056572
- [Derived] Bendabenda J, Patson N, Hallamaa L, Ashorn U, Dewey KG, Ashorn P, Maleta K. Does anthropometric status at 6 months predict the over-dispersion of malaria infections in children aged 6-18 months? A prospective cohort study. Malar J. 2019 Apr 22;18(1):143. doi: 10.1186/s12936-019-2778-y. PMID 31010435
- [Derived] Bendabenda J, Patson N, Hallamaa L, Mbotwa J, Mangani C, Phuka J, Prado EL, Cheung YB, Ashorn U, Dewey KG, Ashorn P, Maleta K. The association of malaria morbidity with linear growth, hemoglobin, iron status, and development in young Malawian children: a prospective cohort study. BMC Pediatr. 2018 Dec 28;18(1):396. doi: 10.1186/s12887-018-1378-2. PMID 30593271
- [Derived] Kumwenda C, Hemsworth J, Phuka J, Ashorn U, Arimond M, Maleta K, Prado EL, Haskell MJ, Dewey KG, Ashorn P. Association between breast milk intake at 9-10 months of age and growth and development among Malawian young children. Matern Child Nutr. 2018 Jul;14(3):e12582. doi: 10.1111/mcn.12582. Epub 2018 Jan 19. PMID 29349922
- [Derived] Adams KP, Ayifah E, Phiri TE, Mridha MK, Adu-Afarwuah S, Arimond M, Arnold CD, Cummins J, Hussain S, Kumwenda C, Matias SL, Ashorn U, Lartey A, Maleta KM, Vosti SA, Dewey KG. Maternal and Child Supplementation with Lipid-Based Nutrient Supplements, but Not Child Supplementation Alone, Decreases Self-Reported Household Food Insecurity in Some Settings. J Nutr. 2017 Dec;147(12):2309-2318. doi: 10.3945/jn.117.257386. Epub 2017 Oct 4. PMID 28978680
- [Derived] Prado EL, Abbeddou S, Adu-Afarwuah S, Arimond M, Ashorn P, Ashorn U, Brown KH, Hess SY, Lartey A, Maleta K, Ocansey E, Ouedraogo JB, Phuka J, Some JW, Vosti SA, Yakes Jimenez E, Dewey KG. Linear Growth and Child Development in Burkina Faso, Ghana, and Malawi. Pediatrics. 2016 Aug;138(2):e20154698. doi: 10.1542/peds.2015-4698. PMID 27474016
- [Derived] Bendabenda J, Alho L, Ashorn U, Cheung YB, Dewey KG, Vosti SA, Phuka J, Maleta K, Ashorn P. The effect of providing lipid-based nutrient supplements on morbidity in rural Malawian infants and young children: a randomized controlled trial. Public Health Nutr. 2016 Jul;19(10):1893-903. doi: 10.1017/S1368980016000331. Epub 2016 Mar 9. PMID 26956611
- [Derived] Hemsworth J, Kumwenda C, Arimond M, Maleta K, Phuka J, Rehman AM, Vosti SA, Ashorn U, Filteau S, Dewey KG, Ashorn P, Ferguson EL. Lipid-Based Nutrient Supplements Increase Energy and Macronutrient Intakes from Complementary Food among Malawian Infants. J Nutr. 2016 Feb;146(2):326-34. doi: 10.3945/jn.115.215327. Epub 2016 Jan 6. PMID 26740684
- [Derived] Maleta KM, Phuka J, Alho L, Cheung YB, Dewey KG, Ashorn U, Phiri N, Phiri TE, Vosti SA, Zeilani M, Kumwenda C, Bendabenda J, Pulakka A, Ashorn P. Provision of 10-40 g/d Lipid-Based Nutrient Supplements from 6 to 18 Months of Age Does Not Prevent Linear Growth Faltering in Malawi. J Nutr. 2015 Aug;145(8):1909-15. doi: 10.3945/jn.114.208181. Epub 2015 Jun 10. PMID 26063066
- [Derived] Ashorn U, Alho L, Arimond M, Dewey KG, Maleta K, Phiri N, Phuka J, Vosti SA, Zeilani M, Ashorn P. Malawian Mothers Consider Lipid-Based Nutrient Supplements Acceptable for Children throughout a 1-Year Intervention, but Deviation from User Recommendations Is Common. J Nutr. 2015 Jul;145(7):1588-95. doi: 10.3945/jn.114.209593. Epub 2015 May 20. PMID 25995276
- [Derived] Kumwenda C, Dewey KG, Hemsworth J, Ashorn P, Maleta K, Haskell MJ. Lipid-based nutrient supplements do not decrease breast milk intake of Malawian infants. Am J Clin Nutr. 2014 Mar;99(3):617-23. doi: 10.3945/ajcn.113.076588. Epub 2013 Dec 24. PMID 24368436
- See also: College of Medicine homepage — http://www.medcol.mw/